CLINICAL TRIAL: NCT00637286
Title: A Multicenter, Open-Label Study Using the MIDAS Questionnaire to Assess the Effect of Using the HCPC Guidelines for Migraine Management in Primary Care, Including the Use of Zomig-ZMT (Zolmitriptan) Orally Disintegrating Tablets 5.0mg and Zomig Nasal Spray 5.0mg as Indicated.
Brief Title: ZAP, US. Zomig for Appropriate for Primary Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1223C00002
Record Dates: First submitted 2008-02-08; First posted 2008-03-17 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-04

CONDITIONS: Migraine
Keywords: Zolmitriptan; ZOMIG; migraine; headache response; headache; headache pain; MIDAS; HCPC
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — zolmitriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Zolmitriptan — 5mg Nasal Spray
  Other Names: Zomig

SUMMARY:
The purpose of this study is to determine how useful and effective the use of ZOMIG-ZMT™ (zolmitriptan) 5.0 mg and ZOMIG® Nasal Spray (zolmitriptan) 5.0 mg is for patients, in treating migraine over a period of 6 months

ELIGIBILITY:
Inclusion Criteria:

* Have an established diagnose of migraine as with an age at onset of less than 50 years
* Have experienced an average of at least 1 migraine headache per month in the previous three months
* Be able to differentiate between migraine and non-migraine headaches

Exclusion Criteria:

* Use of any triptan within the last 12 months or use of MAO-A inhibitors, methysergide or methylergonovine in the 2 weeks before entering the study.
* History of basilar, ophthalmoplegic or hemiplegic migraine headache or any potentially serious neurological condition that is associated with headache
* History, symptoms, or significant risk factors for ischaemic heart or other cardiovascular disease, including coronary vasospasm, cardiac accessory conduction pathways or arrhythmias or uncontrolled hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-07; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Change in Migraine Disability Assessment questionnaire (MIDAS) score | Twice within 28 weeks

SECONDARY OUTCOMES:
Explore patients assessment of value of zolmitriptan | Maximum of 3 times between 1 - 28 weeks